CLINICAL TRIAL: NCT02855671
Title: The Application of Infrared Thermal Imaging in the Diagnosis and Prognostication of Septic Illness in Adults
Brief Title: Infrared Imaging in Septic Illness
Status: Completed | Type: Observational
Sponsor: University Hospitals, Leicester (Other)
Collaborators: Association of Anaesthetists of Great Britain and Ireland (Unknown)
Responsible Party: Sponsor
Other Study IDs: UHL 11486
Record Dates: First submitted 2016-06-20; First posted 2016-08-04 (Estimated); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Sepsis
Keywords: microcirculation; thermal; temperature
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- Healthy volunteers
  Interventions: Device: Infrared thermal imaging
- Sepsis
  Interventions: Device: Infrared thermal imaging
- Severe sepsis/septic shock
  Interventions: Device: Infrared thermal imaging

INTERVENTIONS:
Device: Infrared thermal imaging — Patients in all groups will undergo infrared thermal imaging of the face and anterior leg (centered on the knee)

SUMMARY:
The application of infrared thermal imaging in the diagnosis and prognostication of septic illness in adults.

During times of severe infection (sepsis), the small blood vessels supplying oxygen and nutrients to the skin and other organs (called the microcirculation), become abnormal and do not function as they normally would in health. Monitoring these small blood vessels is difficult to do clinically and the investigators want to investigate a new way of doing this.

The aim of this study is to validate a novel method of assessing the function of the microcirculation in healthy volunteers and patients with sepsis, by measuring the skin temperature profile of the leg and face with a thermal imaging camera. Thermal imaging cameras measure the heat given off by all objects and represents this as a picture, with colour used to represent the different temperatures.

Patients will be recruited from the Emergency Department and Intensive Care Units at University Hospitals of Leicester in to one of two groups based on their illness severity; uncomplicated sepsis and severe sepsis. Healthy volunteers will be recruited in to a third group. Recruitment will take place over a 6-month period with follow-up lasting for 12-months following recruitment. 105 participants will be recruited in total.

Temperature patterns seen on the face and leg will be investigated between the different groups. Changes in these temperature patterns as patients recover from sepsis (or indeed become worse), will also be investigated. Information from the thermal images will be correlated to routinely measured markers of infection, including clinical measurements (blood pressure, pulse, etc) and routine blood investigations.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged 18 years or above.
2. Healthy volunteers - free from acute illness; will include staff and students at the University of Leicester and UHL, and patient relatives.
3. Patient with septic illness will be recruited in to one of two groups depending on their disease severity - Sepsis (without evidence of organ dysfunction) or severe sepsis (with organ dysfunction).
4. Able (in the Investigators opinion) and willing to comply with all study requirements.

Exclusion Criteria:

1. Patient refusal
2. Inability to gain appropriate assent/consent
3. Children
4. Prisoners or in police custody
5. Skin marking likely to preclude image analysis (such as extensive tattoos).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will involve the recruitment of acutely unwell patients from the Emergency Department and Intensive Care Unit areas of the hospital, alongside healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2016-07; Primary Completion 2019-02-01 (Actual); Study Completion 2019-02-01 (Actual)

PRIMARY OUTCOMES:
Measure the extent of thermally apparent mottling of the anterior knee using a previously described mottling score. | 18 months
  Measure the extent of mottling (graded from 1 to 5) using the mottling score described by Ait-Oufella et al.
Measure core-peripheral temperature difference by means of a facial thermal image (Thermal Core-Peripheral Temperature Difference - TCPTD). | 18 months
  Thermal core-peripheral temperature difference (TCPTD) will be assessed using temperature at the medial canthus (core) and nasal (peripheral) in degrees centigrade.

SECONDARY OUTCOMES:
Association between the severity of thermally derived mottling score and the Sequential Organ Failure Assessment (SOFA) score. | 18 months
  Association between mottling score (graded 1-5) and illness severity as determined by the SOFA score (0-24).
Association between the severity of thermally derived mottling score and the APACHE II score. | 18 months
  Association between mottling score (1-5) and illness severity as determined by the APACHE II score (0-71).
Association between the extent of Thermal Core Peripheral Temperature Difference (TCPTD) and the SOFA score. | 18 months
  Associations between TCPTD (degrees centigrade) and illness severity as determined by the SOFA score (0-24).
Association between the extent of Thermal Core Peripheral Temperature Difference (TCPTD) and the APACHE II score. | 18 months
  Associations between TCPTD (degrees centigrade) and illness severity as determined by the APACHE II score (0-71).
Mortality at 30 days and 1 year from the point of enrollment. | 18 months
  Mortality information will be collected at 30 days and 1 year from the point of patient enrollment (0-6 months) and correlated to the thermally derived mottling score and thermal core-peripheral temperature difference to assess for potential prognostic value of the above investigations.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Thompson, MB ChB, BSc, MD, Principal Investigator — University Hospitals, Leicester
Locations (1):
- University Hospitals of Leicester, Leicester, Leicestershire, United Kingdom